CLINICAL TRIAL: NCT00970112
Title: O Uso de Dexametasona e Etoricoxibe Para a prevenção e Controle da Dor pós-operatória após Cirurgia Periodontal
Brief Title: Dexamethasone and Etoricoxib for Pain Prevention Following Periodontal Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Responsible Party: Gibson Luiz Pilatti, UEPG
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08169/08; 51/2008
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-03

CONDITIONS: Pain Control
Keywords: pain; pain assessment
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo 1 hour before surgery
  Interventions: Procedure: Open Flap Debridement
- Etoricoxib (Experimental): Etoricoxib 1 hour before surgery
  Interventions: Procedure: Open Flap Debridement
- Dexamethaone (Experimental): Dexamethasone 1 hour before surgery
  Interventions: Procedure: Open Flap Debridement

INTERVENTIONS:
Procedure: Open Flap Debridement — Open flap debridement - access flap + scaling and root planning

SUMMARY:
The purpose of this study is to investigate whether preemptive medication with dexamethasone or etoricoxib provides better pain management and control than placebo following periodontal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting moderate or severe periodontitis after nonsurgical periodontal treatment with clinical signs of inflammation

Exclusion Criteria:

* Pregnant
* Diabetes mellitus
* Heart diseases
* Allergic to components of the medications
* Risk of endocarditis

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
pain | up to 3 days
  hourly for the 8 first hours after surgery 3 times a day on the following 3 days

CONTACTS AND LOCATIONS:
Overall Officials: João Paulo Steffens, MSc Student, Principal Investigator — UEPG; Fábio André Santos, PhD, Study Director — UEPG; Gibson Luiz Pilatti, PhD, Study Chair — UEPG
Locations (1):
- UEPG, Ponta Grossa, Paraná, Brazil